CLINICAL TRIAL: NCT01846247
Title: A Phase 3, Multicentre, Randomised Controlled Trial of Very Early Rehabilitation After Stroke.
Brief Title: A Very Early Rehabilitation Trial
Acronym: AVERT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuroscience Trials Australia (Other)
Collaborators: Singhealth Foundation (Other Government); Chest, Heart and Stroke Association Scotland (Other); Northern Ireland Chest Heart and Stroke (Other); The Stroke Association - UK (Unknown); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: version3 25April08; ACTRN12606000185561 (Registry Identifier: ANZCTR)
Record Dates: First submitted 2013-04-30; First posted 2013-05-03 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Stroke
Keywords: stroke
MeSH Terms: conditions — Stroke | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Care (Placebo Comparator): Standard stroke unit rehabilitation care
  Interventions: Other: Standard care
- Standard Care + VEM (Experimental): Standard stroke unit rehabilitation care in addition to a very early rehabilitation protocol
  Interventions: Other: Standard Care + VEM

INTERVENTIONS:
Other: Standard Care + VEM — Patient will receive standard stroke unit care with earlier and additional physiotherapy and nursing sessions as per an intervention protocol.
  Arms: Standard Care + VEM
Other: Standard care
  Arms: Standard Care

SUMMARY:
Phase 3, multicenter, international randomized controlled trial of a Very Early Mobilization(VEM) care rehabilitation protocol compared to standard post stroke care (SC). Participants receive either SC and VEM or SC alone in the acute phase of stroke up to a period of 14 days.

Participants are followed up by a blinded assessor at 3 and 12 months post stroke to determine trial outcomes.

DETAILED DESCRIPTION:
People who suffer a stroke are often left with disabilities such as weakness, or problems with speech, thinking, or control or bodily functions. Severe strokes often result in death. The results of a recent European study indicated that patients who commence mobility training very early after a stroke (Day 1) recover the ability to walk more quickly and return home sooner and in greater numbers than those who start training one week or later after stroke. Recently a phase II (pilot) AVERT study was conducted in which the investigators tested the safety and feasibility of very early mobilisation (European model) Stroke patients in this study randomly received either standard care or very early mobilisation (VEM). The study showed that there was no harm to patients in the VEM group compared to those who had standard care and that delivering VEM was feasible. Consequently, a grant to conduct the larger phase III study, to test the effectiveness of the intervention was obtained.

In this next phase III trial, the investigators aim to look at 2104 patients across stroke care units in city and regional hospitals. Each hospital will be asked to include between 30 and 60 patients per year to the study. All stroke patients admitted to the hospital Stroke Unit or ward at the hospital will be invited to participate. Medical clearance will be obtained for all potential participants. Those unconscious or too ill, together with those already participating in acute drug trials will be excluded. Patients who are able will provide their own consent to participate. Those who are not able to consent for themselves will have a third party (usually a relative) acknowledge their participation in the study. As this is a blinded controlled trial, keeping the assessor and patients unaware of their treatment group is important. The investigators will inform patients that they will have a 50% chance of receiving one of two rehabilitation types during their hospitalization if they decide to participate. Patients in the VEM group will commence treatment within 24 hours of admission to hospital. VEM will be provided by a trained AVERT physiotherapist, and AVERT study nurse and aims to improve functional mobility. The mobilization activities will depend on the patient's functional ability and tolerance to exercise. Patients will be closely monitored prior to mobilization and will only be mobilised if they meet requirements for blood pressure and other vital signs. The number of sessions and the time spent for each patient will vary, however specific targets are to be met according to the intervention protocol. The content and timing of all treatment received by participants in either group will be recorded. The treatment period for this study is from the time of the patients consent, until day 14 or discharge from the stroke unit or ward. (Whichever is earlier). All participants will be assessed at admission to the study, 3 months, and 12 months after their stroke. Information collected by the AVERT physiotherapists and nurses and the assessor will be recorded on individual case record forms and on a secure web based data base. Therapists also add some information to a palm pilot, and then download it onto the secure website. All information collected from patients will be treated as confidential in line with international guidelines and local law.

The primary outcome measure for the study is the number of patients dead and disabled at 3 months after stroke. Other secondary outcome measures include the safety of patients, quality of life, and cost effectiveness. An independent Data Monitoring committee will monitor the safety, conduct and efficacy of the trial. In addition, an independent outcomes committee will be reviewing all events that are reported as serious.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Clinical diagnosis of first or recurrent stroke, hemorrhage or infarct.
* Recruited within 24 hours of onset of stroke symptoms
* Admission in a stroke care unit
* Consciousness: At a minimum patient must at least react to verbal commands.

Exclusion Criteria:

* pre stroke mRS of 3,4 or 5
* Deterioration in patients condition resulting in direct admission to ICU, decision to palliate or surgery.
* Concurrent diagnosis of rapidly deteriorating disease
* Unstable coronary or other medical condition that is judged by the investigator to impose a hazard to the patient by involvement
* Patients unable to be mobilized within 24 hours of onset. (eg bed rest policy post tPA, lower limb fracture)
* Other interventional trials
* Systolic BP less than 110 or greater than 220mmHg
* Oxygen saturation of less than 92 % with supplementation
* Resting heart rate of less than 40 or greater than 110 beats per minute
* Temperature of greater than 38.5 degrees C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2014 (Estimated)
Dates: Start 2006-06; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
modified Rankin Score | 3 months
  Favorable outcome (0-2) modified Rankin Score

SECONDARY OUTCOMES:
Safety. Death rate and severity of important medical events | up until 3 months
  Important medical events (stroke progression, recurrent stroke, falls, angina, myocardial infarction, deep vein thrombosis, pulmonary emboli, pressure sores, chest infections, urinary tract infections, depression) at 3 months.
Time to unassisted walking over 50 meters and the proportion achieving unassisted walking | 3 Months
  Achieves walking independently or with supervision over 50 meters
modified Rankin Score | 3 months
  Assumption free ordinal approach
Health related Quality of life | 12 months
  AQoL
Cost effectiveness and cost utility | 12 months
  comprehensive questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Julie Bernhardt, PhD, Study Director — The Florey Institute of Neuroscience and Mental Health; Leonid Churilov, PhD, Principal Investigator — The Florey Institute of Neuroscience and Mental Health; Helen Dewey, MD, Principal Investigator — Monash University; Richard Lindley Dewey, MD, Principal Investigator — George Institute for Global Health; Janice Collier, PhD, Principal Investigator — The Florey Institute of Neuroscience and Mental Health; Amanda Thrift, PhD, Principal Investigator — Monash University; Geoffrey Donnan, MD, Principal Investigator — The Florey Institute of Neuroscience and Mental Health
Locations (1):
- Florey Institute for Neuroscience and Mental health, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Saunders DH, Mead GE, Fitzsimons C, Kelly P, van Wijck F, Verschuren O, Backx K, English C. Interventions for reducing sedentary behaviour in people with stroke. Cochrane Database Syst Rev. 2021 Jun 29;6(6):CD012996. doi: 10.1002/14651858.CD012996.pub2. PMID 34184251
- [Derived] Sheppard L, Dewey H, Bernhardt J, Collier JM, Ellery F, Churilov L, Tay-Teo K, Wu O, Moodie M; AVERT Trial Collaboration Group. Economic Evaluation Plan (EEP) for A Very Early Rehabilitation Trial (AVERT): An international trial to compare the costs and cost-effectiveness of commencing out of bed standing and walking training (very early mobilization) within 24 h of stroke onset with usual stroke unit care. Int J Stroke. 2016 Jun;11(4):492-4. doi: 10.1177/1747493016632254. Epub 2016 Mar 2. PMID 26936861
- [Derived] Bernhardt J, Raffelt A, Churilov L, Lindley RI, Speare S, Ancliffe J, Katijjahbe MA, Hameed S, Lennon S, McRae A, Tan D, Quiney J, Williamson HC, Collier J, Dewey HM, Donnan GA, Langhorne P, Thrift AG; AVERT Trialists' Collaboration. Exploring threats to generalisability in a large international rehabilitation trial (AVERT). BMJ Open. 2015 Aug 17;5(8):e008378. doi: 10.1136/bmjopen-2015-008378. PMID 26283667